CLINICAL TRIAL: NCT02632799
Title: Airway Pressure During Nasal High Flow and CPAP in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Center of Maternal and Child Health Protection, Armenia (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RCMCHP012
Record Dates: First submitted 2015-09-10; First posted 2015-12-17 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Respiratory Insufficiency
Keywords: Nasal High Flow; CPAP; airway pressure; newborn
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- NHF small cannula (Experimental): NHF 8 L/min (Airvo2) , Smaller cannula (neonatal, yellow)
  Interventions: Device: NHF small cannula
- NHF big cannula (Experimental): NHF 8 L/min (Airvo2) , Bigger cannula (neonatal, purple)
  Interventions: Device: NHF big cannula
- Mask CPAP (Experimental): CPAP 5cm H2O
  Interventions: Device: CPAP
- no intervention (No Intervention): control

INTERVENTIONS:
Device: NHF small cannula — NHF 8 l/min by Airvo 2 by small cannula
  Other Names: Optiflow, HFNC
  Arms: NHF small cannula
Device: NHF big cannula — NHF 8 l/min by Airvo 2 by large cannula
  Other Names: Optiflow, HFNC
  Arms: NHF big cannula
Device: CPAP — Nsal CPAP 5cm H2o by face mask
  Arms: Mask CPAP

SUMMARY:
Nasal High Flow (NHF) and CPAP are established forms of respiratory support in neonates and often produce similar clinical outcomes. The aim of the study was to investigate airway pressure during NHF and CPAP in neonates.

DETAILED DESCRIPTION:
Methods: A physiological study which measured pressure intra-nasally with micro (750 µm) pressure probes (Millar, USA) in 10 (5M / 5F) healthy newborns with mean gestation age 37.18 (SD 1.29) wk and mean birth weight of 2414 (SD 503.13) g. NHF was applied at 8 L/min (AIRVO 2) through smaller (OPT 314) and larger (OPT 316) Optiflow nasal cannula; CPAP 5 cmH20 was produced by a Bubble CPAP system and nasal mask interface at constant flow 8 L/min (Fisher & Paykel Healthcare, NZ). Values are expressed in cmH20 as means and standard deviations (SD).

ELIGIBILITY:
Inclusion Criteria:

* Healthy term newborns

Exclusion Criteria:

* Newborns with any medical problems after birth
* Absent of parents consents

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Upper airway pressure generated by NHF compared to CPAP | Up to 1 hour
  Pressure in upper airways

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Mazmanyan, MD PhD, Principal Investigator — Research Center of Maternal and Child Health Protection, Armenia
Locations (2):
- Armenia (2):
  - Neonatal Intensive Care Unit, Research Centre of Maternal and Child Health, Yerevan
  - RCMCHP, Yerevan